CLINICAL TRIAL: NCT06937125
Title: Evaluation of Valvular Heart Disease: Multicenter Registry of Noninvasive Imaging Modalities by Cardiac CT
Brief Title: Evaluation of Valvular Heart Disease Using Cardiac CT
Status: Recruiting | Type: Observational
Sponsor: Toho University (Other)
Responsible Party: Principal Investigator, Hideki Koike, Principal Investigator, Toho University
Other Study IDs: A24904
Record Dates: First submitted 2025-04-18; First posted 2025-04-22 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The EVIDENTIA Registry is a multicenter study designed to evaluate valvular heart disease (VHD) using cardiac CT. It aims to assess cardiac valve anatomy, function, and myocardial characteristics through detailed CT analysis.

1. Assessing the accuracy of cardiac CT in evaluating cardiac structure, volume, function, and myocardium in VHD patients.
2. Comparing the severity, classification, and etiology (primary vs. functional) of VHD.
3. Monitoring serial changes in VHD severity via echocardiography.
4. Investigating the relationship between echocardiographic and CT-derived parameters.
5. Examining the correlation between imaging findings, VHD interventions, and patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least moderate valvular heart disease who had a cardiac CT with 64 or more rows
* 18 years of age or older

Exclusion Criteria:

* Less than 18 years old
* Acute VHD
* Infectious endocarditis
* Patients with post-VHD intervention
* Poor CT image quality for analyzing CT data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at 7 centers throughout Japan, with the goal of enrolling a total of approximately 300-350 cases.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
the 1-year composite endpoint of all-cause death and major cardiac adverse events (MACE) including VHD intervention. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Toho University, Ōta-ku, Tokyo, Japan